CLINICAL TRIAL: NCT06917092
Title: A Phase II Study to Evaluate the Efficacy and Safety of QL1706 Combination Therapy in Immunotherapy-Pretreated Recurrent or Metastatic Endometrial Cancer
Brief Title: QL1706-Based Therapy Post-PD-1/L1 Failure in Advanced Endometrial Cancer
Acronym: QLPPEC/GOG-003
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: E20250167
Record Dates: First submitted 2025-04-01; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Endometrial Adenocarcinoma; Endometrial Cancer
Keywords: Immunotherapy-Pretreated; Recurrent or Metastatic Endometrial Carcinoma; Immune Checkpoint Inhibitors; QL1706
MeSH Terms: conditions — Endometrial Neoplasms; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QL1706 Combination Therapy (Experimental): QL1706 Combination Therapy in Immunotherapy-Pretreated Recurrent or Metastatic Endometrial Carcinoma
  Interventions: Drug: QL1706 combined with chemotherapy ± Bevacizumab

INTERVENTIONS:
Drug: QL1706 combined with chemotherapy ± Bevacizumab — * Drug: QL1706: 5 mg/kg IV every 3 weeks until progression, unacceptable toxicity, completion of 1 year of treatment, or meeting protocol-defined discontinuation criteria, whichever occurred first.
  * Drug: Chemotherapy: physician's choice chemotherapy for 3-6 cycles.
  * Drug: Bevacizumab (optional): 15 mg/kg IV every 3 weeks until progression, unacceptable toxicity, completion of 1 year of treatment, or meeting protocol-defined discontinuation criteria, whichever occurred first.

SUMMARY:
This is a prospective, single-arm, multicenter Phase II study evaluating the efficacy and safety of QL1706 combined with chemotherapy in patients with advanced recurrent or metastatic endometrial cancer who progressed after prior anti-PD-1/L1 therapy.

DETAILED DESCRIPTION:
This prospective, single-arm, multicenter Phase II study evaluates the efficacy and safety of QL1706 plus physician's choice chemotherapy (with or without bevacizumab) in patients with advanced recurrent or metastatic endometrial cancer refractory to prior PD-1/L1 inhibitor therapy. The study consists of three phases: screening, treatment, and post-treatment follow-up, with continuous safety monitoring throughout. Eligible patients had confirmed disease progression following previous PD-1/L1 inhibitor treatment. Participants received QL1706 combined with physician's choice chemotherapy, with or without bevacizumab. All participants will undergo post-treatment safety monitoring and survival follow-up after treatment completion. For patients who discontinue treatment for reasons other than disease progression or death, additional tumor progression follow-up will be conducted post-treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years and ≤70 years.
2. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
3. Recurrent or metastatic endometrial carcinoma, confirmed by pathology or imaging.
4. At least one measurable tumor lesion according to RECIST v1.1 criteria.
5. Patients must have received prior anti-PD-1/L1 monoclonal antibody (mAb) therapy with a progression-free survival (PFS) of ≥6 months; however, the last dose of anti-PD-1/L1 mAb must have been administered at least 5 half-lives before the initiation of the current treatment.
6. Patients who have received prior anti-angiogenic therapy are eligible, provided there is a washout period of at least 5 half-lives before re-administration.
7. Patients who have failed ≤2 lines of prior systemic therapy are eligible (endocrine therapy is not counted as a line of treatment).
8. All other anti-tumor therapies must be discontinued at least 4 weeks before treatment initiation. Patients taking hormonal medications require a 30-day washout period.
9. Laboratory tests during the screening period must demonstrate adequate organ function.
10. Female subjects of childbearing potential must have a negative serum pregnancy test within 3 days prior to the first dose. If a female subject of childbearing potential engages in sexual activity with a non-sterilized male partner, the subject must use an acceptable and highly effective contraceptive method since screening and must agree to continue such precautions until 6 months after the last dose of the study drug; periodic abstinence and the rhythm method are not acceptable forms of contraception.
11. Voluntarily sign the informed consent form, understand the nature, purpose, and procedures of the trial, and willingly comply with the trial requirements.

Exclusion Criteria:

* 1. Previous treatment with PD-1/CTLA-4 dual-target immunotherapy, immune checkpoint agonists (e.g., ICOS, CD40, CD137, GITR, OX40 antibodies, etc.), or immune cell therapy.

  2. Discontinuation of anti-PD-1/PD-L1 antibody therapy due to related toxicity. 3. Presence of any active autoimmune disease or history of autoimmune disease (including but not limited to autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hypophysitis, vasculitis, nephritis, hyperthyroidism; patients with vitiligo or childhood asthma that has completely resolved and requires no intervention in adulthood may be included; asthma requiring bronchodilator treatment is excluded).

  4. Current use of immunosuppressants or systemic corticosteroids for immunosuppression (dose >10 mg/day prednisone or equivalent) within 2 weeks prior to enrollment.

  5. Known active tuberculosis (TB) or suspected active TB requiring clinical evaluation for exclusion; known active syphilis infection.

  6. History of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.

  7. History of severe allergic reactions to monoclonal antibodies. 8. Known history or evidence of interstitial lung disease or active non-infectious pneumonitis.

  9. History or current presence of central nervous system (CNS) metastases. Baseline imaging to confirm the absence of brain metastases is not mandatory. Patients with unknown CNS status but clinical signs suggestive of CNS metastases must be excluded via CT/MRI.

  10. History of other malignancies (except non-melanoma skin cancer or cervical carcinoma in situ; patients with other prior malignancies must have been disease-free for at least 3 years).

  11. Uncontrolled hypertension despite antihypertensive therapy (systolic BP ≥140 mmHg or diastolic BP ≥90 mmHg); hypertensive crisis or hypertensive encephalopathy in the past.

  12. History of unstable angina, myocardial infarction (MI), chronic heart failure (CHF), clinically significant arrhythmias requiring treatment (except stable atrial fibrillation), or left ventricular ejection fraction <50% within 6 months before the first dose.

  13. Current thrombolytic or anticoagulant therapy (prophylactic low-dose aspirin or low molecular weight heparin is permitted).

  14. Arterial/venous thrombotic events within 6 months before enrollment (e.g., cerebrovascular accident, transient ischemic attack, cerebral hemorrhage, cerebral infarction, deep vein thrombosis, pulmonary embolism).

  15. Major vascular disease within 6 months before study treatment (e.g., aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis).

  16. Major surgery within 4 weeks before study treatment (excluding diagnostic procedures) or anticipated major surgery during the study.

  17. Prior radiotherapy (except palliative bone radiotherapy), chemotherapy, or surgery (excluding biopsy) within 4 weeks before the first study dose; last antibody dose <4 weeks before study treatment; molecular targeted therapy (including other investigational oral targeted agents) <5 half-lives before study treatment; or unresolved toxicities (>CTCAE grade 1, except alopecia) from prior therapy.

  18. Active infection, unexplained fever ≥38.5°C within 7 days before treatment, or baseline white blood cell count >15×10⁹/L.

  19. Congenital or acquired immunodeficiency (e.g., HIV infection); HBsAg-positive with HBV DNA ≥2000 IU/mL, or HCV antibody-positive.

  20. Live/attenuated vaccination within 4 weeks before study treatment or anticipated during the study.

  21. Any other condition deemed by the investigator to potentially affect study results or lead to premature termination.

  22. Pregnant or breastfeeding women.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) - Investigator assessment | Up to 5 years
  the objective response rate (ORR) of treatment with QL1706 combined with chemotherapy ± Bevacizumab, as assessed by the Investigator per RECIST v.1.1.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) - investigator assessment | Up to 5 years
  the Progression-Free Survival (PFS) of treatment with QL1706 combined with chemotherapy ± Bevacizumab, as assessed by the Investigator per RECIST v.1.1.
Overall survival (OS) | Up to 5 years
  the overall survival (OS) of treatment with QL1706 combined with chemotherapy ± Bevacizumab, as assessed by the Investigator per RECIST v.1.1.
Duration of response (DOR) - Investigator assessment | Up to 5 years
  the duration of response (DOR) of treatment with QL1706 combined with chemotherapy ± Bevacizumab, as assessed by the Investigator per RECIST v.1.1.
Number of participants with adverse events (AEs), Serious adverse events (SAEs) and treatment-emergent adverse events (TEAEs) | Up to 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute & Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No